CLINICAL TRIAL: NCT05839080
Title: FoodACT: Investigating the Impact of a School Garden Intervention on Children's Food Literacy, Climate Literacy, Physical Activity, and School Motivation
Brief Title: FoodACT: Investigating the Impact of a School Garden Intervention on Children's Food Literacy, Climate Literacy, School Motivation and Physical Activity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Clinical Research and Prevention (Network)
Collaborators: University of Copenhagen (Other); Haver til Maver (Unknown)
Responsible Party: Principal Investigator, Peter Elsborg, Principal Investigator, Center for Clinical Research and Prevention
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NFF22SH0077522
Record Dates: First submitted 2023-03-10; First posted 2023-05-03 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-09

CONDITIONS: Physical Inactivity; Literacy; Motivation
Keywords: School; Physical activity; Outdoor; School garden; Motivation; Food literacy; Climate literacy; Education; Health Promotion
MeSH Terms: conditions — Sedentary Behavior; Literacy; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study has two different participant samples. In Sub-Study 1 the participants are pupils from 4th-5th grade from Danish municipal primary and lower secondary schools attending the 'Gardens to Bellis' intervention (intervention group) and pupils from 4th-5th grade from Danish municipal primary and lower secondary schools not attending the 'Gardens to Bellis' intervention.
  In Sub-Study 2 and Sub-Study 3, the participant sample is a subsample of the intervention sample in SS1. The participants are pupil's 4th-5th grade (n=540) from 30 Danish municipal primary and lower secondary schools.
Masking Description: It is not possible to mask the participants since they are signed up for the Gardens to Bellis intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention schools (Experimental): Pupils are exposed to the schoolgarden intervention eight times during two school years
  Interventions: Behavioral: Gardens to Bellis
- Control Schools (Experimental): Pupils are not exposed to the interventions and will complete questionaries
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: Gardens to Bellis — In FoodACT the school garden intervention that will be investigated is the well described and well-developed intervention called Gardens to Bellis. It involves pupils from 4th-5th grade and their teachers. The classes attend 8 school garden sessions distributed across two school years. The sessions start each year in March and ends in November. Pupils are divided into smaller groups, who gets a plot of which they are responsible for preparing, weed and harvest. The purpose is that pupils can cook their own food with the greens, fruits and berries they harvest in the garden and finds in the nature. The pupils and their families will hatch and harvest the school gardens between the session days.
  Other Names: FoodACT
  Arms: Intervention schools
Behavioral: No intervention — Pupils are not receiving any intervention
  Arms: Control Schools

SUMMARY:
The purpose of this study is to investigate the efficacy of a schoolgarden intervention on pupils food literacy, climate literacy, schoolmotivation and physical activity. The study will also investigate the contextual characteristics in the garden using systematic observations and the pupil´s experience of the intervention with focus-groups interviews.

DETAILED DESCRIPTION:
Globally, the prevalence of obesity and severe obesity among children and youth is rising. Inactivity and unhealthy diet are often associated with obesity which can lead to detrimental health outcomes such as cardiovascular disease and type-2 diabetes. Schools are considered a key setting for promoting children and adolescents' food literacy, climate literacy, physical activity and to improve their mental and social health. Interventions in schools have a broad impact because all children spent the majority of their waking hours in school independent of their socio-economic- and cultural background. FoodACT aims to invetigate an well-established schoolgarden intervention on pupils food literacy, climate literacy, schoolmotivation and physical activity.

School gardens create an enabling environment for increasing student's food literacy and climate literacy, where an active component is that the pupils cultivate and prepare their own crops through a program that extends through nine months and therefore becomes an integrated part of the pupils schooling. The children's' physical activty is affected without it being the focus of the school garden programs. Pupils get up from the chair in the classroom, use active transportation for example by foot or bike to the school garden and are activated by work such as digging, lifting and watering their own plot. Some school garden interventions also invovle and activate the pupils families, which increases the sustainability of the interventions effects. Previous research has stated that schools are considered a key setting for promoting children and adolescents' food literacy and physical activity and to improve their mental and social health. Relocating teaching to an outdoor nature setting, which is a central ingredients of school garden interventions, has shown to be positively related to increased physical activity in both boys and girls during the school day. Furthermore, contextual and experience related characteristics such as tasks, motions, associations and interactions realted to the school garden has not been captured.

Therefore, the aim of FoodACT is to investigate how a school gardening intervention impact pupils food literacy, climate literacy, school motivation and physical activity with a special focus on children with low socio-economics in a controlled design.

In 2023 a pilot-study will be performed to test and adjust the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* 4th-5th grade school classes in Danish municipal primary and lower secondary schools participating in the 'Gardens to Bellis' intervention.
* Classes not involved in other school development or research projects.
* Participants with parents (or legal guardian) having provided written informed consent.

Exclusion Criteria:

• Pupils with significant health problems as judged by the investigators will be excluded from the analysis (Sub-study 1-3).

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 990 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity (PA) | 9 months
  Physical activity will be measured with Sens Motion accelerometers or with Axivity® AX3 accelerometer as described above. The primary outcomes are pupils' physical activity i.e., sedentary behaviour (SED), light physical activity (LPA), moderate-to-vigorous physical activity (MVPA).
  Using Sens motion all acceleration data will be processed and transferred into a secure web server via the smartphone. Based on the sensor's orientation (axes) and acceleration, a predefined algorithm categorises the measurements in predefined behaviour activities, e.g., sitting, lying down, standing, walking, cycling and number of steps. In addition, a categorisation of intensity levels is predefined e.g., moderate, and high physical activity.
Food literacy (FL) | 9 months
  FL will be measured using the Food Literacy Quesionare designed for school children (FLQ-sc; (Stjernqvist, Elsborg, et al., 2021). The questionnaire is developed and validate to school children in 6th and 7th grade (aged 12-14). It's a 37 item questionnaire used to access individual FL which is based on Benn 2014 five FL competencies: "to know, "to do", "to sense", "to care" and "to want".
  Measured two times in 2024 where change is being assesed.
Climate Literacy (CL) | 9 months
  CL will be measured based on a Climate Litercy Quesionare (Dewaters et.al. 2011), which will be modified and adapted during the pilot-study targeting the right age-group.
  Measured two times in 2024 where change is being assesed.
School motivation (SM) | 9 months
  School motivation (SM) will be measured using the Academic Self-Regulation Questionnaire (called SRQ-A). The SRQ-A is a domain-specific self-report questionnaire developed for measuring the level of autonomy relative to doing different types of schoolwork among pupils in late primary and lower-secondary school.
  Measured two times in 2024 where change is being assesed.

SECONDARY OUTCOMES:
Systematic observations with PARAGON | 9 months
  The primary outcomes are the pupil's movements, postures, motions, and experience of the intervention activities. When using systematic observations with PARAGON (The Physical Activity Research and Assessment tool for Garden Observation) pupils' movements and motions will be captured when they attend the gardening intervention activities. The observed movements and motions are categorised into four categories: overall PA-level, garden-related tasks, garden related motions, social associations, and interaction
Focus-group interviews | 9 months
  Semi-structured focus-group interviews will be held after a day with gardening intervention activities with both the involved pupils, teachers, parents (or legal guardian) and gardens facilitators. The thematic content analyses will be open to unforeseen themes that may emerge while also keeping a focus on the different target groups' motivation and experience with the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Research and Prevention, Frederiksberg, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant-level data can be made available upon reasonable request to the PI such as e.g. verification of the research results. To comply with the European General Data Protection Regulation, and to accommodate article 10 of the Danish Act on Data Protection anonymised participant-level data will be made available on the Open Science Framework five years after the main publication of this study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Anonymised participant-level data will be made available on the Open Science Framework five years after the main publication of this study.
  Statistical plan, study protocol and analytical code will be made available in the osf folder upon acceptance of first preregistered manuscript.
Access Criteria: Data can be made available upon reasonable request to the PI such as e.g. verification of the research results.

REFERENCES:
- [Derived] Stage A, Vermund MC, Bolling M, Otte CR, Oest Mullertz AL, Bentsen P, Nielsen G, Elsborg P. The impact of a school garden program on children's food literacy, climate change literacy, school motivation, and physical activity: A study protocol. PLoS One. 2025 Apr 24;20(4):e0320574. doi: 10.1371/journal.pone.0320574. eCollection 2025. PMID 40273231
- See also: FoodACT website — http://www.foodact.dk